CLINICAL TRIAL: NCT06639165
Title: Retrospective-perspective Observational Cohort Study on Toxicity and Efficacy of Radiotherapy in Pediatric and Adult Patients With Pediatric Histology Treated at the Pediatric Radiotherapy of the CRO in Aviano
Acronym: RADIOPED
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2020-65
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Radiation Toxicity
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiotherapy key role in pediatric oncology, despite the potential side effects especially in the long term, including the risk of radioinduced second cancers.

Very rarely malignant neoplasms typical of children and adolescents may present in adulthood, historically with a worse outcome, but for some of these histologies demonstrated recent results overlapping with those in pediatric age when treated with strategies similar to pediatric protocols and similar radiotherapy.

Long-term data on outcome and incidence of potential toxicity late radiation therapy in these populations almost exclusively from epidemiologic studies or retrospective case series. Prospective data are lacking, particularly in patients treated with IMRT and specifically with certain IMRT modalities such as Helical Tomotherapy, for which the CRO pediatric radiotherapy has documented experience. The main objective is to evaluate the short- and long-term toxicity secondary to radiotherapy performed at the Pediatric Radiotherapy of the CRO in Aviano, with specific subgroup analyses aimed at highlighting any differences mainly by age, pathology and radiotherapy technique.

DETAILED DESCRIPTION:
Radiotherapy key role in pediatric oncology, despite the potential side effects especially in the long term, including the risk of radioinduced second cancers.

Very rarely malignant neoplasms typical of children and adolescents may present in adulthood, historically with a worse outcome, but for some of these histologies demonstrated recent results overlapping with those in pediatric age when treated with strategies similar to pediatric protocols and similar radiotherapy.

Long-term data on outcome and incidence of potential toxicity late radiation therapy in these populations almost exclusively from epidemiologic studies or retrospective case series. Prospective data are lacking, particularly in patients treated with IMRT and specifically with certain IMRT modalities such as Helical Tomotherapy, for which the CRO pediatric radiotherapy has documented experience.

The main objective is to evaluate the short- and long-term toxicity secondary to radiotherapy performed at the Pediatric Radiotherapy of the CRO in Aviano, with specific subgroup analyses aimed at highlighting any differences mainly by age, pathology and radiotherapy technique.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric, adolescent, and young adult (<25 years old) patients with malignant neoplasm
* Adult patients (≥25 years) with malignant neoplasm with histology typical of pediatric age but rarely also found in adults and typically treated wherever possible in pediatric protocols (mainly: Central nervous system malignancies such as medulloblastomas and other embryonal tumors, ependymomas, and germ cell tumors; soft tissue and bone sarcomas such as rhabdomyosarcomas and Ewing's sarcomas; nephroblastomas; neuroblastomas)
* Underwent radiation treatment at the Pediatric Radiotherapy Unit of the CRO in Aviano
* Between October 24, 1991, and September 30, 2020, with regard to the retrospective phase of the study, and between October 1, 2020, and September 30, 2030, with regard to the prospective phase of the study
* And who provide informed consent to the study if alive and traceable at the time of enrollment with regard to the retrospective phase of the study and necessarily with regard to the prospective phase. Regarding deceased or alive but untraceable patients enrollable in the retrospective phase of the study, since these are patients who had already given consent to data processing at the time of the radiation therapy being analyzed and registration/enrollment in any specific treatment/research protocols, no new consent is required for the study

Exclusion Criteria:

- Anything not covered in the inclusion criteria

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All pediatric, adolescent and young adult (<25 years old) patients with malignant neoplasm e All adult patients (≥25 years) with malignant neoplasm with histology typical of pediatric age but also rarely found in adults and typically treated wherever possible in pediatric protocols (mainly: malignant tumors affecting the central nervous system such as medulloblastomas and other embryonal tumors, ependymomas, and tumors with germ cells; soft tissue and bone sarcomas such as rhabdomyosarcomas and Ewing's sarcomas; nephroblastomas; neuroblastomas) undergoing radiation treatment at the pediatric radiation therapy of the CRO of Aviano
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute radiotherapy-related side effects | up to 10 years
  Cumulative incidence of acute side effects, with degree of individual toxicities encountered defined according to the most up-to-date version of the Common Terminology Criteria for Adverse Events (CTCAE) available at the time of analysis; analysis by subgroups of patients.
Incidence of chronic side effects related to radiotherapy | up to 10 years
  Cumulative incidence of chronic side effects, with degree of the individual toxicities encountered defined according to the most up-to-date version of the CTCAE available at the time of analysis; analysis by subgroups of patients
Incidence of second cancers | up to 10 years
  Cumulative incidence of second cancers; analysis by subgroups of patients.

SECONDARY OUTCOMES:
Patient survival in terms of overall survival (OS, overall survival) and progression-free survival (PFS, progression-free survival) | up to 10 years
  Data will be summarized with survival curves according to Kaplan-Meier method; differences between selected subgroups of patients will be assessed by log-rank test. OS will be defined as time from beginning of the therapy until death from any cause or end of follow-up, whichever comes first.
Adequacy of radiation treatment understood as compliance with the requirements in terms of target coverage | up to 10 years
  Frequency of patient with adequate target coverage
Adequacy of radiation treatment understood as dose conformation to the target | up to 10 years
  Frequency of patient with adequate dose conformation to the target selection of alternative plans deemed superior and/or developed retrospectively with new radiotherapy techniques not yet available at the initial planning stage; qualitative-quantitative dosimetric comparisons between plans
Homogeneity of dose to the target | up to 10 years
  Frequency of patient with homogeneity of dose to the target

CONTACTS AND LOCATIONS:
Locations (1):
- Centro di Riferimento Oncologico, Aviano, Pordenone, Italy